CLINICAL TRIAL: NCT02896270
Title: A Prospective Interventional Pilot Study on the Use of Valproic Acid for Treatment of Idiopathic Nephrotic Syndrome
Brief Title: Valproic Acid for Idiopathic Nephrotic Syndrome
Acronym: VAIN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UZB_20160728
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Idiopathic Nephrotic Syndrome; Focal Segmental Glomerulosclerosis; Minimal Change Disease
Keywords: idiopathic podocytopathies; Neprology
MeSH Terms: conditions — Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): Patients will start study treatment on Day1 and will be treated with a dose of 250mg twice daily of the valproic acid slow release formulation (Depakine Chrono© - Sanofi Pharma Belgium).
  Control of valproic acid serum levels after 4 to 7 days. The dose will be progressively increased targeting valproic acid serum levels in the target range for use of the drug as an anti-epileptic (50-100µg/ml).
  During the study, visits will be performed every month and at the end of treatment. The duration of the study is 12 months. Continuation of valproic acid after completion of the study will be at the investigators discretion.
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid — The concomitant immunosuppressive regimen is to be reduced at the discretion of the investigators. It is suggested to lower immunosuppressive therapy only in valproic acid target trough levels have been attained.
  Other Names: Depakine Chrono 500©, Sanofi

SUMMARY:
The trial investigates the use of VPA (Valproic Acid) for the treatment of adult patients with biopsy proven idiopathic focal segmentel glomerulosclerosis (FSGS) or minimal change disease (MCD).

VPA used as an add-on to steroids might induce clinical remission in a first category of patients and potentially reduce the dose of maintenance immunosuppression required to maintain remission thereafter.

In a second category of patients VPA might allow the reduction or even cessation of immunosuppression while clinical remission is maintained.

DETAILED DESCRIPTION:
Idiopathic MCD to treat diseases with a considerable associated morbidity and mortality. Current treatment options are limited, have limited efficacy and a considerable side effect profile. Recent findings in a murine model suggest that VPA treatment in an early phase of renal disease could halt or even prevent the development of proteinuria and the progression of kidney damage. VPA is a commonly used and easy available oral antiepileptic agent with a favorable side effect profile compared to the current standard of care agents for podocytopathies.

This trial investigates wether

1. VPA on top of or in substitution of standard of care agents is effective in remission induction in patients with FSGS or MCD with proteinuria resistant to first line therapy with corticosteroids.
2. VPA is effective in remission maintenance allowing reduction and cessation of chronic immunosuppression without relapse in patients with frequently relapsing FSGS or MCD.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Biopsy proven idiopathic FSGS or MCD
* Organ function:

  * Bilirubin/AST/ALT< 2 ULN
  * PLT>100.000 10*6/L
  * INR 1.5 except if on anti-vitamin K treatment
  * Lipase <1.5 ULN
  * Creatinine clearance >30ml/min -

Exclusion Criteria:

* Contraindication for VPA
* Secondary etiologies for FSGS or MCD
* Multiple organ transplantation
* Currently participating in another clinical trial
* Pregnant or lactating women
* Women unwilling to take efficient contraceptive measures for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
In remission group induction is the proportion of patients in complete remission | 6 months
  Complete remission is defined as a reduction of proteinuria to <300mg/g creatinine or < 0.3g/d and normal serum creatinine (or stable creatinine if baseline creatinine before disease onset is well documented) and serum albumin > 3.5g/dL.
In remission maintenance group is the proportion of patients able to reduce maintenance | 6 months
  The proportion of patients able to reduce maintenance immunosuppression to a monotherapy of 4 mg methylprednisolone or less while remaining in complete remission

SECONDARY OUTCOMES:
Determine the disease response by the proportion of subjects with partial remission | 6 - 12 months
  Remission induction patients with partial remission defined as a reduction in proteinuria to 0.3-3.5g/d or 300-3500mg/g creatinine and a decrease of at least 50% from baseline proteinuria and stable serum creatinine (change in creatinine < 25%) 6 months after inclusion into the study for FSGS.
  Remission maintenance patients remaining in remission for at least 6 months after reduction of maintenance immunosuppression to monotherapy with 4 mg of methylprednisolone or less.
Determine the extent to which standard immunosuppression can be reduced | 6 - 12 months
  The proportion of "remission induction patients" attaining full or partial remission with 4mg methylprednisolone or less 6 months and 12 months after inclusion; The proportion of "remission maintenance patients" remaining in remission for at least 6 months after reduction of maintenance immunosuppression to monotherapy with 4 mg of methylprednisolone or less.
Evaluate the evolution of renal function estimated by MDRD-GFR | 12 months
  Evolution of renal function estimated by CKD-EPI
Evaluate the tolerability of VPA in the setting of idiopathic podocytopathies | 12 months
  Evaluation adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Peter Janssens, MD, Principal Investigator — University Hospital Brussels, Belgium
Locations (2):
- Belgium (2):
  - University Hospital Brussels, Brussels
  - UVC Brugmann, Brussels

IPD SHARING:
Plan to Share IPD: Yes
The data of this pilot study will be submitted for publication as soon as the anticipated 15 subjects have completed the study.